CLINICAL TRIAL: NCT02200471
Title: Evaluation of VeinViewer in Cosmetic Dermatology
Brief Title: Cosmetic Dermatology Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christie Medical Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: SPN - 13 / 04 - 01
Record Dates: First submitted 2014-07-21; First posted 2014-07-25 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Cosmetic Procedures
Keywords: Cosmetic dermatology; near-infrared; patient preference; physician preference
MeSH Terms: conditions — Patient Preference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- VeinViewer (Experimental): VeinViewer will be used in conjunction with routine cosmetic dermatology procedures. Patients and physicians will complete questionnaires.
  Interventions: Device: VeinViewer

INTERVENTIONS:
Device: VeinViewer

SUMMARY:
This study aims to understand the impact of VeinViewer technology during routine cosmetic and dermatologic procedures.

DETAILED DESCRIPTION:
This study was designed as an observational study to determine if VeinViewer technology helped to improve the efficiency of certain dermatological procedures namely botox injections and schlerotherapy for varicose veins. The device was used to identify veins but clinical decisions were ultimately left the physician.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and up
* Male or Female
* Receiving cosmetic dermatological injection
* Willing to participate

Exclusion Criteria:

* Aged younger than 18 years
* Prior history of known light sensitivity
* Other reasons as determined by investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2013-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Patient perception of the use of the device | Day 1
  Small questionnaires will be used to assess how the patient perceives the use of the device (i.e., did the patient have a positive attitude towards the device?)

SECONDARY OUTCOMES:
Physician perception of the use of the device | Day 1
  Physicians will complete a small questionnaire to understand what their perception of the use of the device to be (i.e, did the physician have a positive attitude towards the device while using it).

OTHER OUTCOMES:
Detection of adverse events related to the standard of care procedure | 2nd day
  VeinViewer may be used to detect adverse events related to the standard of care procedure (e.g., bruising).

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dermatology Cosmetic Laser Medical Associates of La Jolla, Inc., La Jolla, California
  - MD Laser Skin & Vein Institute, Hunt Valley, Maryland